CLINICAL TRIAL: NCT02300116
Title: Smart Vision Labs Autorefractor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Smart Vision Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: 28/OCT/2014
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Ocular Refraction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The study is used to verify the accuracy and repeatability of Smart Vision Labs Refractor.

ELIGIBILITY:
Inclusion Criteria:

* healthy young adults
* ages 18-35 year
* male and female

Exclusion Criteria:

* presence of ocular disease
* refractive surgery
* amblyopia

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young adults: ages 18-35 year, including male and female
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
refractive errors | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ciuffreda, O.D, PH.D, Principal Investigator — State University of New York College of Optometry
Locations (1):
- SUNY/College of Optometry, New York, New York, United States